CLINICAL TRIAL: NCT02671526
Title: Plasticity-based Adaptive Cognitive Remediation (PACR) for HIV-associated Neurocognitive Dysfunction
Brief Title: Cognitive Remediation for HIV-associated Neurocognitive Dysfunction
Acronym: HAND
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Posit Science Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PSC-1005-14
Record Dates: First submitted 2016-01-27; First posted 2016-02-02 (Estimated); Last update posted 2016-11-23 (Estimated); Status verified 2016-11

CONDITIONS: HIV-associated Neurocognitive Dysfunction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Computerized Plasticity-based Adaptive Cognitive Training (Experimental)
  Interventions: Other: Computerized plasticity-based adaptive cognitive training

INTERVENTIONS:
Other: Computerized plasticity-based adaptive cognitive training

SUMMARY:
This study is a validation study to document the acceptability of the revised Plasticity-based Adaptive Cognitive Remediation (PACR) program to patients with HIV-associated Neurocognitive Dysfunction (HAND). The primary objective of this study is to evaluate the effects of the revised PACR program on the cognitive abilities (e.g., attention, executive function), functional status and quality of life of individuals diagnosed with HAND. The secondary objective of the study is to collect relevant data to support a pre-investigational device exemption (IDE) submission to the FDA required before the pivotal randomized, controlled trial planned for Phase II.

ELIGIBILITY:
1. Participant is between 25-60 years of age
2. Participant is HIV positive
3. Participant has diagnosis of HIV-associated neurocognitive disorder (HAND), Mild Neurocognitive Disorder (MND) and HIV associated dementia (HAD)
4. Participant is fluent in English
5. Participant is able to use an iPad and have access to wireless internet connection
6. Participant does not have a history of other conditions (other that from HAND), including mental illness, cancer, or other neurological conditions (multiple sclerosis, seizure disorder)
7. Participant is not enrolled in another research study
8. Participant does not have current or significant past history of substance abuse
9. Participant does not have severe depression or other chronic psychiatric disorder (eg. Schizophrenia or Bipolar Disorder)

Ages: 25 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 19 (Actual)
Dates: Start 2015-12; Primary Completion 2016-11 (Actual); Study Completion 2016-11 (Actual)

PRIMARY OUTCOMES:
Computerized Exercise-based Assessment | 3 months
  The primary outcome measure is the useful field of view; change on this measure suggests underlying neural change, and has been shown to predict overall cognitive change. The exercise-based measure serves as a positive control for task learning. The investigators anticipate improvements in this assessment because participants have directly practiced these tasks, as well as tasks within related cognitive domains. The data are relevant because individuals failing to make progress on this assessment may represent a subpopulation not treatable with this program, and individuals making strong progress may represent a subpopulation particularly amenable to treatment with this program. This assessment will be performed on the first day of program use, approximately halfway through program use, and the last day of program use. All participants will access this assessment via Internet portal and study team member may access results via clinician portal.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas Van Vleet, Ph.D., Principal Investigator — Posit Science Corporation
Locations (1):
- Posit Science Corporation, San Francisco, California, United States